CLINICAL TRIAL: NCT03075865
Title: The OmniMax MMF System: A Cohort Study for Clinical Evaluation
Brief Title: A Cohort Study for Clinical Evaluation of OmniMax MMF System
Acronym: OmniMax
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Collaborators: University of Iowa (Other); Medical University of South Carolina (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1116
Record Dates: First submitted 2017-03-03; First posted 2017-03-09 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Mandibular Fractures
Keywords: intermaxillary fixation; maxillo-mandibular fixation
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- OmniMax MMF: Patients involved in trauma events will receive intermaxillary fixation with OmniMax MMF system for temporary stabilization of mandibular fracture(s) to maintain proper occlusion during surgery and allow for postoperative fracture healing.
  Interventions: Device: OmniMax MMF system

INTERVENTIONS:
Device: OmniMax MMF system — OmniMax MMF system consists of arch bars and screws that work together to achieve temporary fixation of the maxilla and mandible to provide indirect or passive stabilization of fractures and maintenance of occlusion in the oral and maxillofacial region. The arch bars have hooks designed to accommodate either wires or elastic bands for temporary maxillomandibular fixation (MMF) either intraoperative or postoperative.
  Other Names: OmniMax

SUMMARY:
OmniMax MMF system was designed as a device with faster application/removal time, less mucosal tissue overgrowth over the plates and screws, better tolerance for placement over prolong periods of time, better patient hygiene and a lower risk for further treatments secondary to root damage from the insertion of the screws, compared to the standard of care for maxillo-mandibular fixation and other hybrid systems. This clinical trial intends to highlight the clinical benefits of the OmniMax MMF system applied to patients undergoing repair of uncomplicated mandibular fracture(s) for whom OmniMax MMF system is used as a single mean for maxillo-mandibular fixation.

DETAILED DESCRIPTION:
The objective of this study is to highlight and evaluate the clinical benefits of OmniMax MMF system applied to patients undergoing repair of uncomplicated mandibular fracture(s). A total of 50 subjects involved in trauma events resulting in uncomplicated mandibular fracture(s) will be enrolled at up to 5 sites from 3 surgical subspecialties: maxillofacial surgery, ENT, and plastic surgery. Subjects considered for participation will receive OmniMax MMF system for maxillo-mandibular fixation for a period of 4 to 8 weeks. Incidence of root damage associated with screw insertion, time for implantation and removal of the device, oral hygiene during the maxillomandibular fixation period, mucosal overgrowth, gingival necrosis, post-operative pain, stability of the occlusion, fracture healing, patient overall satisfaction/compliance with length of treatment, incidence of glove perforation and accidental puncture, will be evaluated in all participants who remain in IMF post-operatively. Adverse Events associated with the use of OmniMax MMF system will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* 18 years of age or older
* Able and willing to sign ICF and medical photography consent
* Undergoing a surgical procedure to repair uncomplicated mandibular fracture(s) requiring open reduction internal fixation (ORIF) or closed maxillo-mandibular fixation (MMF)
* Fracture repair done within 10 days after facial trauma
* Use of OmniMax MMF system as a single mean for IMF (maxillary plate and mandibular plates together with no other device combined, such as Erich bars or IMF screws).

Exclusion Criteria:

* General contraindications unfavorable for the use of MMF (psychological disorders, seizures disorders, airway compromise, immune-compromised patients, etc).
* History of radiation therapy to the head or neck region.
* Limited blood supply to the area of device application.
* Insufficient quantity or quality of bone.
* History of foreign body sensitivity.
* History of previous use of bisphosphonates (i.e. alendronate, pamidronate, neridronate, olpadronate, ibandronate, risendronate, zolendronate).
* Clinically active or latent infection.
* Patients with less than 20 teeth.
* Deciduous dentition.
* Patients for whom the use of OmniMax MMF system would not be appropriate in judgment of the surgeon (i.e., excessive overjet or deep overbite).
* Mandibular fracture pattern that could prevent the use of OmniMax MMF system for adequate reduction and stabilization (i.e., comminuted fractures, dental alveolar fractures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults involved in trauma events resulting in uncomplicated mandibular fractures and needing intermaxillary fixation for fracture repair and fracture healing.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Root Damage | 6 weeks
  Dental root damage can be caused from insertion of the screws at time of implantation. Some of these events may require further medical or surgical treatment

SECONDARY OUTCOMES:
Time for Implantation of OmniMax MMF | Operative
  The OmniMax MMF system, with a better segmentalized design and extended screw slots, allows for fixation of this device using less quantity of screws for fixation (compared to other hybrid systems). This system may impact the efficiency of the medical care by significantly reducing the operative time.
Tissue necrosis and mucosal overgrowth | 6 weeks
  The reduced number of screws needed to fixate a full OmniMax MMF system (8 versus up to 14 in other bone-borne systems) is expected to improve the post-operative gingival tissue health, avoiding soft tissue irritation, overgrowth, compression and necrosis of the gingival area.

OTHER OUTCOMES:
Patient Satisfaction | 6 weeks
  Less screws for fixation and design of the device to protect the soft tissue is expected to increase the level of patient satisfaction and patient compliance with both, the oral hygiene and the length of fixation period.
Gloves Perforation and Accidental Puncture | Operative
  Design of OmniMax MMF system is expected to reduce the risk for accidental glove perforation and/or wire puncture during implantation of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Hatcher, PhD, Study Director — Zimmer Biomet CMF & Thoracic
Locations (3):
- United States (3):
  - University of California Davis Medical Center, Sacramento, California
  - University of Iowa, Iowa City, Iowa
  - College of Dental Medicine, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engelstad ME, Kelly P. Embrasure wires for intraoperative maxillomandibular fixation are rapid and effective. J Oral Maxillofac Surg. 2011 Jan;69(1):120-4. doi: 10.1016/j.joms.2010.06.209. Epub 2010 Oct 29. PMID 21035935
- [Background] Ansari K, Hamlar D, Ho V, Hilger P, Cote D, Aziz T. A comparison of anterior vs posterior isolated mandible fractures treated with intermaxillary fixation screws. Arch Facial Plast Surg. 2011 Jul-Aug;13(4):266-70. doi: 10.1001/archfacial.2011.46. PMID 21768561
- [Background] Sahoo NK, Mohan R. IMF Screw: An Ideal Intermaxillary Fixation Device During Open Reduction of Mandibular Fracture. J Maxillofac Oral Surg. 2010 Jun;9(2):170-2. doi: 10.1007/s12663-010-0049-0. Epub 2010 Sep 22. PMID 22190780
- [Background] Cornelius CP, Ehrenfeld M. The Use of MMF Screws: Surgical Technique, Indications, Contraindications, and Common Problems in Review of the Literature. Craniomaxillofac Trauma Reconstr. 2010 Jun;3(2):55-80. doi: 10.1055/s-0030-1254376. PMID 22110819
- [Background] Roccia F, Rossi P, Gallesio C, Boffano P. Self-tapping and self-drilling screws for intermaxillary fixation in management of mandibular fractures. J Craniofac Surg. 2009 Jan;20(1):68-70. doi: 10.1097/SCS.0b013e318190df2f. PMID 19164992
- [Background] Bagheri SC, Dimassi M, Shahriari A, Khan HA, Jo C, Steed MB. Facial trauma coverage among level-1 trauma centers of the United States. J Oral Maxillofac Surg. 2008 May;66(5):963-7. doi: 10.1016/j.joms.2008.01.020. PMID 18423287
- [Background] Gaujac C, Ceccheti MM, Yonezaki F, Garcia IR Jr, Peres MP. Comparative analysis of 2 techniques of double-gloving protection during arch bar placement for intermaxillary fixation. J Oral Maxillofac Surg. 2007 Oct;65(10):1922-5. doi: 10.1016/j.joms.2006.06.311. PMID 17884516
- [Background] Coletti DP, Salama A, Caccamese JF Jr. Application of intermaxillary fixation screws in maxillofacial trauma. J Oral Maxillofac Surg. 2007 Sep;65(9):1746-50. doi: 10.1016/j.joms.2007.04.022. PMID 17719392
- [Background] Fabbroni G, Aabed S, Mizen K, Starr DG. Transalveolar screws and the incidence of dental damage: a prospective study. Int J Oral Maxillofac Surg. 2004 Jul;33(5):442-6. doi: 10.1016/j.ijom.2003.10.014. PMID 15183406
- [Background] Ayoub AF, Rowson J. Comparative assessment of two methods used for interdental immobilization. J Craniomaxillofac Surg. 2003 Jun;31(3):159-61. doi: 10.1016/s1010-5182(03)00022-2. PMID 12818601
- [Background] Vartanian AJ, Alvi A. Bone-screw mandible fixation: an intraoperative alternative to arch bars. Otolaryngol Head Neck Surg. 2000 Dec;123(6):718-21. doi: 10.1067/mhn.2000.111286. PMID 11112964
- [Background] Valentino J, Marentette LJ. Supplemental maxillomandibular fixation with miniplate osteosynthesis. Otolaryngol Head Neck Surg. 1995 Feb;112(2):215-20. doi: 10.1016/S0194-59989570239-3. PMID 7838541
- [Background] Hashemi HM, Parhiz A. Complications using intermaxillary fixation screws. J Oral Maxillofac Surg. 2011 May;69(5):1411-4. doi: 10.1016/j.joms.2010.05.070. Epub 2011 Jan 8. PMID 21216063
- [Background] Nandini GD, Balakrishna R, Rao J. Self Tapping Screws v/s Erich Arch Bar for Inter Maxillary Fixation: A Comparative Clinical Study in the Treatment of Mandibular Fractures. J Maxillofac Oral Surg. 2011 Jun;10(2):127-31. doi: 10.1007/s12663-011-0191-3. Epub 2011 Apr 20. PMID 22654363
- [Background] Rai A, Datarkar A, Borle RM. Are maxillomandibular fixation screws a better option than Erich arch bars in achieving maxillomandibular fixation? A randomized clinical study. J Oral Maxillofac Surg. 2011 Dec;69(12):3015-8. doi: 10.1016/j.joms.2010.12.015. Epub 2011 Apr 5. PMID 21470746
- [Background] Schulte-Geers M, Kater W, Seeberger R. Root trauma and tooth loss through the application of pre-drilled transgingival fixation screws. J Craniomaxillofac Surg. 2012 Oct;40(7):e214-7. doi: 10.1016/j.jcms.2011.10.022. Epub 2011 Nov 17. PMID 22099624
- [Background] Park KN, Oh SM, Lee CY, Kim JY, Yang BE. Design and application of hybrid maxillomandibular fixation for facial bone fractures. J Craniofac Surg. 2013;24(5):1801-5. doi: 10.1097/SCS.0b013e3182a21163. PMID 24036784
- [Background] Chao AH, Hulsen J. Bone-supported arch bars are associated with comparable outcomes to Erich arch bars in the treatment of mandibular fractures with intermaxillary fixation. J Oral Maxillofac Surg. 2015 Feb;73(2):306-13. doi: 10.1016/j.joms.2014.08.025. Epub 2014 Aug 27. PMID 25488313
- [Background] Ingole PD, Garg A, Shenoi SR, Badjate SJ, Budhraja N. Comparison of intermaxillary fixation screw versus eyelet interdental wiring for intermaxillary fixation in minimally displaced mandibular fracture: a randomized clinical study. J Oral Maxillofac Surg. 2014 May;72(5):958.e1-7. doi: 10.1016/j.joms.2014.01.005. Epub 2014 Jan 18. PMID 24642133
- [Background] West GH, Griggs JA, Chandran R, Precheur HV, Buchanan W, Caloss R. Treatment outcomes with the use of maxillomandibular fixation screws in the management of mandible fractures. J Oral Maxillofac Surg. 2014 Jan;72(1):112-20. doi: 10.1016/j.joms.2013.08.001. Epub 2013 Sep 25. PMID 24075236
- [Background] Meursinge Reynders R, Ladu L, Ronchi L, Di Girolamo N, de Lange J, Roberts N, Pluddemann A. Insertion torque recordings for the diagnosis of contact between orthodontic mini-implants and dental roots: protocol for a systematic review. Syst Rev. 2015 Apr 2;4:39. doi: 10.1186/s13643-015-0014-6. PMID 25875916
- [Background] Laurentjoye M, Majoufre-Lefebvre C, Siberchicot F, Ricard AS. Result of maxillomandibular fixation using intraoral cortical bone screws for condylar fractures of the mandible. J Oral Maxillofac Surg. 2009 Apr;67(4):767-70. doi: 10.1016/j.joms.2008.06.055. PMID 19304032